CLINICAL TRIAL: NCT02372721
Title: Long Term Impact of Pediatric Acute Renal Injury in Severe Sepsis
Acronym: IMPRESS
Status: Withdrawn | Type: Observational
Why Stopped: The IRB required this protocol to be split into two different protocols
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400925
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease; Hypertension
Keywords: acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sepsis with Severe AKI: History of a pediatric admission with sepsis related AKI which lead to classification of "injury" or "failure". This group will have urinary and serum studies to measure glomerular filtration rate, renal plasma flow followed by cardiovascular assessments using blood pressure monitoring, peripheral arterial and applanation tonometry.
- Sepsis without AKI: History of a pediatric admission with sepsis which lead to no classification of AKI. This group will have urinary and serum studies to measure glomerular filtration rate, renal plasma flow followed by cardiovascular assessments using blood pressure monitoring, peripheral arterial and applanation tonometry.
- Control: No history of an admission for AKI. This group will have urinary and serum studies to measure glomerular filtration rate, renal plasma flow followed by cardiovascular assessments using blood pressure monitoring, peripheral arterial and applanation tonometry.

SUMMARY:
Sepsis is the most common cause of childhood death worldwide. Millions of children survive, but are left with impaired health. Sepsis-related Acute Kidney Injury (sAKI) is increasingly recognized as a significant factor associated with long-term mortality among different patient populations. Renal dysfunction and subsequent chronic kidney disease is implicated in the development of hypertension and cardiovascular disease. The investigators overall hypothesis is that, in the pediatric population, sepsis-related AKI will have unrecognized, long-term consequences with regard to kidney function, endothelial function, blood pressure control, and overall health.

DETAILED DESCRIPTION:
This will be a three-arm cross-sectional control-cohort outpatient evaluation. Subjects with sAKI and a random selection of non-sAKI subjects who agree to participate in another study of quality of life survey will be asked to participate in the outpatient study. Subjects will be asked to come in to the Clinical Research Center for 24-hour monitoring and participate in the outpatient study where urinary and serum studies to measure glomerular filtration rate, renal plasma flow followed by blood pressure monitoring, peripheral arterial and applanation tonometry.

ELIGIBILITY:
Inclusion Criteria:

For non-acute kidney injury (AKI) sepsis patients:

1. Hospitalization with a diagnosis of sepsis from 1998-2014
2. Failure to meet pediatric Risk Injury Failure Loss End stage (pRIFLE) criteria for AKI during incident admission.
3. Participation in cognitive survey study with completion of survey

For sepsis related AKI patients:

1. Hospitalization with a diagnosis of sepsis from 1998-2014
2. Need for renal replacement therapy (RRT)
3. Severe AKI as defined by the pRIFLE criteria (estimated CrCl (eCrCl) decrease by 50%, eCrCl <60 ml/min/1.73 m2, or a urine output <0.5 ml/kg/h for 24 h or anuric for 12 h) during the sepsis admission
4. Participation in cognitive survey study with completion of survey

For healthy control patients:

1. Identified from the neurology service who are scheduled for MRI with gadolinium as part of their clinical care

Exclusion Criteria:

For all patients:

1. Known pre-existing chronic kidney disease (CKD) as defined by history of kidney transplant or long-term dialysis
2. Age greater than 18 years at the time of sepsis admission
3. AKI from primary kidney disease including acute glomerulonephritis and obstructive uropathy
4. Pregnancy at the time of enrollment
5. Age younger than 5, between the ages of 12 to 17, or over the age of 24 at the time of enrollment.

For healthy control patients:

1. Chronic kidney injury (CKD)
2. History of acute kidney injury
3. History of any chronic illnesses (e.g. cancer)

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We intend to contact and enroll patients with severe sepsis related AKI patients without sepsis related AKI and a sample of age and sex-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Chronic Kidney Disease | Day 2
  Obtaining preliminary estimates of glomerular function, renal plasma flow, proteinuria, cystatin C and microalbuminuria in children with and without a history of acute kidney injury in order to assess the presence of chronic kidney disease.

SECONDARY OUTCOMES:
Hypertension | 24 hours
  Ambulatory blood pressure (BP) monitoring, peripheral arterial and applanation tonometry will be performed. A subject will be considered hypertensive if systolic and/or diastolic blood pressure is >95th percentile for sex, age, and height.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Carmelle Elie, MD, Principal Investigator — University of Florida